CLINICAL TRIAL: NCT01074099
Title: Feasibility Study of Autologous Concentrated Bone Marrow Nucleated Cell Therapy for Congestive Heart Failure Patients Undergoing Treatment With Coronary Artery Bypass Grafting(CABG) Surgery
Brief Title: Feasibility Study of BMAC Enhanced CABG
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Pilot results in change to protocol, new study needed.
Sponsor: Harvest Technologies (Industry)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Harvest 2009-1
Record Dates: First submitted 2010-02-01; First posted 2010-02-24 (Estimated); Results first posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2014-08

CONDITIONS: Congestive Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): CABG only
  Interventions: Procedure: CABG only
- BMAC enhanced CABG (Experimental): Injection of concentrated bone marrow nucleated cells (BMAC) as an adjunct to CABG surgery
  Interventions: Biological: BMAC

INTERVENTIONS:
Biological: BMAC — Injection of BMAC into ischemic myocardium during CABG
  Arms: BMAC enhanced CABG
Procedure: CABG only — Control subjects will undergo CABG surgery without BMAC injection
  Arms: Control

SUMMARY:
Patients undergoing CABG will have 60 mL of bone marrow drawn, concentrated in a SmartPRep2 centrifuge and have the concentrated nucleated cells injected into areas of ischemic myocardium

DETAILED DESCRIPTION:
Patients undergoing CABG will have 60 mL of bone marrow drawn, concentrated in a SmartPRep2 centrifuge and have the concentrated nucleated cells injected into areas of ischemic myocardium. Control subjects will undergo CABG only

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years and ability to understand the planned treatment.
* Patients with ischemic congestive heart failure requiring by pass surgery
* Congestive heart failure with ejection fraction ≤ 40%.
* Serum bilirubin, SGOT and SGPT ≤2.5 time the upper level of normal.
* Serum creatinine < 3.0 or no dialysis.
* NYHA performance status ≥ 3.
* Negative pregnancy test (in women with childbearing potential).
* Subject has read and signed the IRB approved Informed Consent form
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000, Creatinine ≤ 3.0 mg / Dl, and/or no dialysis, INR ≤ 1.6 unless on Coumadin, or PTT <1.5 x control (to avoid bleeding complications) Patients on Coumadin will be corrected prior to the procedure and must have an INR<1.6 at the time of randomization/surgery

Exclusion Criteria:

* Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method, or who intend to become pregnant during the tenure of this study.
* History of Prior Radiation Exposure for oncological treatment.
* History of Bone Marrow Disorder (especially NHL, MDS) that prohibit transplantation.
* History of abnormal Bleeding or Clotting.
* History of Liver Cirrhosis.
* Acute Myocardial Infarction < 4 weeks from treatment date.
* Known active malignancy or results outside of normal limits from the following tests: PAP, Chest X-ray, PSA, Mammogram, Hemoccult unless follow-up studies reveal patient to be cancer free.
* Active clinical infection being treated by antibiotics within one week of enrollment
* Terminal renal failure with existing dependence on dialysis
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.
* Unable to have 250cc bone marrow harvested.
* Medical risk that precludes anesthesia or ASA Class 5
* History of ventricular arrhythmia if AICD is not present.
* History of ventricular aneurysm.
* Concurrent surgery such as CABG with valve surgery.
* Minimally Invasive bypass surgery
* Life expectancy <6 months due to concomitant illnesses
* Treatment with immunosuppressant drugs (including Prednisone > 5 mg per day)
* Patients undergoing urgent by pass surgical procedure
* Patients with HGB A1C > 8.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amit Patel, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - The Methodist Hospital, Houston, Texas
  - University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | BMAC Enhanced CABG
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | BMAC Enhanced CABG | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 3 | 5
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Cardiac Status (Classification)
Description: A change in cardiac status as determined by the New York Heart Association (NYHA) or Canadian Cardiovascular Society (CCS) classification evaluation
Time Frame: Through 12 months post treatment
Population: Study was terminated after enrollment of only 5 patients. The data were not analyzed for efficacy.
Arm/Group | Control | BMAC Enhanced CABG
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Safety
Description: as measured by frequency and severity of adverse events
Time Frame: through 1 Year post tx
Measure: Number; unit: participants
Arm/Group | Control | BMAC Enhanced CABG
Number analyzed (Participants) | 2 | 3
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: From time of treatment through 1 year / study termination
Arm/Group | Control | BMAC Enhanced CABG
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=2) | BMAC Enhanced CABG (N=3)
sustained ventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1) — patient had an episode during the investigational procedure when the injection into the heart occurred. recovered without sequelae

LIMITATIONS AND CAVEATS:
The study was terminated early. Only 5 subjects were enrolled and they were followed for a year for safety data only. One efficacy data was collected.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less